CLINICAL TRIAL: NCT00363883
Title: Phase II Study of Oral Suberoylanilide Hydroxamic Acid (SAHA) in Recurrent or Metastatic Transitional Cell Carcinoma of the Urothelium
Brief Title: Vorinostat in Treating Patients With Locally Recurrent or Metastatic Cancer of the Urothelium
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial stopped early for futility
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02844; NCI-2012-02844 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-61 (Other: City of Hope); 6879 (Other: CTEP); N01CM62209 (NIH); P30CA033572 (NIH)
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2015-02-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Localized Transitional Cell Cancer of the Renal Pelvis and Ureter; Metastatic Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Transitional Cell Cancer of the Renal Pelvis and Ureter; Regional Transitional Cell Cancer of the Renal Pelvis and Ureter; Transitional Cell Carcinoma of the Bladder
MeSH Terms: interventions — Vorinostat

ARMS (1):
- Treatment (vorinostat) (Experimental): Patients receive oral vorinostat (SAHA) twice daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This phase II trial is studying how well vorinostat works in treating patients with locally recurrent or metastatic cancer of the urothelium.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine response rate measured by RECIST criteria for SAHA in patients with recurrent or metastatic transitional cell carcinoma of the urothelium.

SECONDARY OBJECTIVES:

I. To determine the time to progression and overall survival for SAHA in patients with recurrent or metastatic transitional cell carcinoma of the urothelium.

II. To provide data on safety and toxicity of SAHA in patients with recurrent or metastatic transitional cell carcinoma of the urothelium.

III. To obtain preliminary data on molecular correlates in tissue, oral mucosa and blood to determine feasibility and clinical efficacy.

OUTLINE: This is a multicenter study.

Patients receive oral vorinostat (SAHA) twice daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood and buccal mucosa collection and tumor biopsies (if accessible) at baseline and periodically during study for correlative studies. Samples are examined by gene expression profiling and immunohistochemistry.

After completion of study treatment, patients are followed for up to 26 weeks.

PROJECTED ACCRUAL: A total of 37 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathological diagnosis of transitional cell carcinoma of the bladder or urothelium with less than 25% component of other cell types such as small cell, neuroendocrine or squamous cell carcinoma; archival tumor tissue must be available for classification and correlates as described in this protocol or otherwise the patient must be willing to undergo biopsy prior to trial entry
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan; patients with boney metastases are allowed to participate in the study provided they also have non-osseous disease that is measurable
* Patients must have recurred or progressed on or subsequent to platinum-based chemotherapy in the adjuvant or advanced setting; patients treated with a second line of chemotherapy may be included provided more than six months elapsed from the completion of the first line of chemotherapy to the start of the second; patients may have had any number of prior intravesical therapies for superficial bladder cancer; patients may also have had one experimental biologic therapy for their metastatic urothelial cancer provided this was not an agent known to act through histone deacetylation or demethylation; these compounds include sodium butyrate, trichostatin A (TSA), trapoxin (TPX), MS-27-275 and depsipeptide
* Life expectancy of greater than 3 months
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* AST (SGOT)/ALT (SGPT) =< 2.5 x institutional upper limit of normal unless there are liver metastases in which case AST/ALT must be =< 5 x the upper limits of institutional normal
* Creatinine =< 1.5 times normal institutional limits OR creatinine clearance >= 40 mL/min/1.73 m^2 for patients with creatinine levels above 1.5 times institutional normal
* Eligibility of patients receiving any medications or substances known to effect or with the potential to effect the activity or pharmacokinetics of SAHA will be determined following review by the principal investigator
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SAHA; these compounds include sodium butyrate, trichostatin A (TSA), trapoxin (TPX), MS-27-275 and depsipeptide
* Prior treatment with more than 2 cytotoxic chemotherapy regimens for urothelial transitional cell cancer
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this stud; breastfeeding should be discontinued if the mother is treated with SAHA
* HIV-positive patients receiving combination antiretroviral therapy are ineligible
* Patients should not have taken valproic acid for at least two weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Quinn, MD, Principal Investigator — University of Southern California, Norris
Locations (1):
- University of Southern California, Norris, Los Angeles, California, United States

REFERENCES:
- [Derived] Quinn DI, Tsao-Wei DD, Twardowski P, Aparicio AM, Frankel P, Chatta G, Wright JJ, Groshen SG, Khoo S, Lenz HJ, Lara PN, Gandara DR, Newman E. Phase II study of the histone deacetylase inhibitor vorinostat (Suberoylanilide Hydroxamic Acid; SAHA) in recurrent or metastatic transitional cell carcinoma of the urothelium - an NCI-CTEP sponsored: California Cancer Consortium trial, NCI 6879. Invest New Drugs. 2021 Jun;39(3):812-820. doi: 10.1007/s10637-020-01038-6. Epub 2021 Jan 6. PMID 33409898

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Vorinostat)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 65 [43 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Response assessed after every 2 cycles (6 weeks) up to 26 weeks
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 14
percentage of patients | 0

2. Secondary Outcome: Overall Survival
Description: Will be estimated using the product-limit method of Kaplan and Meier.
Time Frame: Up to 26 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 14
months | 4.3 [2.1 to 8.3]

3. Secondary Outcome: Progression-free Survial
Description: Will be estimated using the product-limit method of Kaplan and Meier. Progression defined using RECIST v1.0 criteria, at least a 20% increase in the sum of the longest diameter of target lesions, or the appearance of one or more new lesions.
Time Frame: assessed up to 26 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Vorinostat)
Number analyzed (Participants) | 14
months | 1.1 [1.0 to 2.1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 1 year and 5 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Vorinostat)
Serious Adverse Events (participants affected / at risk) | 6/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vorinostat) (N=14)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Disease progression (General disorders) | 2 (2)
Sudden death (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Intraoperative urinary injury (Injury, poisoning and procedural complications) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vorinostat) (N=14)
Hemoglobin decreased (Blood and lymphatic system disorders) | 8 (18)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (6)
Diarrhea (Gastrointestinal disorders) | 4 (8)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 9 (12)
Vomiting (Gastrointestinal disorders) | 5 (8)
Chills (General disorders) | 1 (1)
Disease progression (General disorders) | 6 (6)
Edema limbs (General disorders) | 4 (4)
Fatigue (General disorders) | 11 (24)
Fever (General disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 5 (8)
Aspartate aminotransferase increased (Investigations) | 5 (8)
Bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 9 (27)
Lymphocyte count decreased (Investigations) | 1 (1)
Lymphopenia (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 6 (20)
Weight loss (Investigations) | 4 (6)
Anorexia (Metabolism and nutrition disorders) | 9 (16)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 3 (3)
Blood glucose increased (Metabolism and nutrition disorders) | 6 (8)
Dehydration (Metabolism and nutrition disorders) | 3 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (17)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (5)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 4 (5)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (2)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Taste alteration (Nervous system disorders) | 2 (5)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 2 (3)
Depression (Psychiatric disorders) | 4 (6)
Insomnia (Psychiatric disorders) | 2 (2)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early after the first stage of a two-stage design, allowing for early termination for discouraging results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less